CLINICAL TRIAL: NCT06988423
Title: A Phase 1, Single-Center, Open-Label, Randomized, Single-Dose, 2-Period, Crossover Study to Evaluate the Potential Impact of High-fat Meal on the Pharmacokinetics of CRS3123 200 mg Capsule in Healthy Adult Participants
Brief Title: Evaluation of the Potential Impact of a High-fat Meal on the Pharmacokinetics of CRS3123 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Crestone, Inc (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 24-3123-FE; 75N93019C00056 (DMID 25-0002) (Other Grant/Funding Number: NIAID)
Record Dates: First submitted 2025-05-16; First posted 2025-05-23 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Food Effect in Healthy Participants
MeSH Terms: interventions — REP 3123

STUDY DESIGN:
Intervention Model Description: In each period, participants will receive Treatment A or Treatment B according to the randomization scheme:
  * Treatment A: No food will be allowed from at least 10 hours before dosing until at least 4 hours after dosing.
  * Treatment B: After a supervised overnight fast of at least 10 hours, participants will be served a high-calorie and high-fat breakfast, in compliance with the FDA Guidance for Industry: Assessing the Effects of Food on Drugs in INDs and NDAs - Clinical Pharmacology Considerations (2022). Breakfast will be served approximately 30 minutes prior to CRS3123 administration. Participants will fast for no less than 4 hours after study drug administration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment A: 1 x 200 mg CRS3123 capsule administered under fasting conditions (Experimental): A single 200 mg dose of CRS3123 administered orally as 1 × 200 mg capsule under fasting conditions.
  Interventions: Drug: CRS3123 200 mg capsule
- Treatment B: 1 x 200 mg CRS3123 capsule administered under fed conditions (Experimental): A single 200 mg dose of CRS3123 administered orally as 1 × 200 mg capsule under fed conditions.
  Interventions: Drug: CRS3123 200 mg capsule

INTERVENTIONS:
Drug: CRS3123 200 mg capsule — CRS3123 200 mg capsule given as a single oral dose

SUMMARY:
This study will explore the potential effects of high-fat meal on the plasma pharmacokinetics (PK) of CRS3123 when administered as a single oral dose of 200 mg in healthy adult participants.

DETAILED DESCRIPTION:
This study will assess the impact of a high-calorie and high-fat meal on the plasma pharmacokinetics (PK) of CRS3123 in healthy adult participants when administered as a single oral capsule of 200 mg dose. Pharmacokinetics (PK) of a single dose of CRS3123 200 mg will be studied following administration to healthy participants under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant and non-lactating adults, non-smoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥ 18 and ≤ 64 years of age, with body mass index (BMI) > 18.5 and < 30.0 kg/m2 and body weight ≥ 50.0 kg for males (as assigned at birth) and ≥ 45.0 kg for females (as assigned at birth), at the time of signing the informed consent.
2. Healthy as defined by:

   1. the absence of clinically significant physical or laboratory findings (above Grade 1) and surgery within 4 weeks prior to dosing.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal (GI), renal, hepatic, and metabolic disease.
3. Healthy females (as assigned at birth) of non-childbearing potential must be:

   1. postmenopausal (spontaneous amenorrhea for at least 12 months prior to dosing) with confirmation by documented follicle stimulating hormone (FSH) levels greater than or equal to 40 mIU/mL; or
   2. surgically sterile (bilateral oophorectomy, hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, bilateral salpingectomy, hysterectomy or tubal ligation) at least 3 months prior to dosing.
4. Sexually active females (as assigned at birth) of childbearing potential and non-sterile males (as assigned at birth) must be willing to use an acceptable contraceptive method throughout the study.
5. Able to understand the study procedures and provide signed informed consent to participate in the study.

Exclusion Criteria:

1. Any clinically significant abnormal finding at physical examination at screening that may interfere with the interpretation of safety and PK objectives of the study.
2. Abnormal laboratory test results (above Grade 1) that may interfere with the interpretation of safety and PK objectives of the study.
3. Positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) antigen and antibody.
4. History of current or chronic liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
5. Positive pregnancy test at screening or admission to the clinical research unit.
6. Positive urine drug screen, urine cotinine test, or alcohol test at screening or admission to the clinical research unit.
7. Known allergic reactions to CRS3123 or other related drugs, or to any excipient in the formulation.
8. Use of medications within specified timeframes.
9. Previous exposure to CRS3123 within 12 months prior to the first dose.
10. Participants with HR < 50 or > 100 beats per minute (bpm), systolic blood pressure (SBP) < 90 or > 140 mmHg, diastolic blood pressure (DBP) < 50 or > 90 mmHg, on vital sign assessment at screening or admission to the clinical research unit.
11. A baseline ECG at screening with corrected QT interval (QTc) using Fridericia's formula (QTcF) > 450 msec.
12. Evidence of previous myocardial infarction (does not include ST segment changes associated with repolarization). Any clinically significant (above Grade 1) conduction abnormality (including but not specific to left or right complete bundle branch block, atrioventricular block [second degree or higher], Wolf Parkinson White syndrome), sinus pauses > 3 seconds, non sustained or sustained ventricular tachycardia (≥ 3 consecutive ventricular ectopic beats) or any significant arrhythmia which, in the opinion of the Investigator will interfere with the safety of the individual participant.
13. Participant has any surgical or medical condition (active or chronic) or GI tract condition (e.g., surgical resection of significant proportions of the stomach or bowel, gastric bypass, gastric banding, irritable bowel syndrome, inflammatory bowel disease, or any other condition that may interfere with normal gastric emptying or transit time) that may interfere with drug absorption, distribution, metabolism, or excretion of the study drug, or any other condition that may place the participant at risk, in the opinion of the Investigator.
14. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days or 5× t½ (whichever is longer) prior to the first dose, administration of a biological product in the context of a clinical research study within 90 days or 5× t½ (whichever is longer) prior to the first dose or concomitant participation in an investigational study involving no drug or device administration.
15. Participants with serum creatinine level > 1.5 mg/dL.
16. History of drug abuse within 1 year prior to screening or recreational use of soft drugs (such as marijuana) within 1 month or hard drugs (such as cocaine, phencyclidine [PCP], crack, opioid derivatives including heroin, and amphetamine derivatives) within 3 months prior to screening.
17. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 10 units for women or 15 units for men of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
18. Donation of plasma within 7 days prior to dosing or donation or loss of 500 mL or more of whole blood within 8 weeks prior to first dosing.
19. Participant is unable to comply with all the study procedures in the opinion of the Investigator.
20. Any reason the participant should not participate in the study in the opinion of the Investigator.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Calculation of AUC0-t for CRS3123 under fasted conditions | 24 hours
  Area under the concentration-time curve from time zero until the last observed concentration under fasted conditions
Calculation of AUC0-t for CRS3123 under fed conditions | 24 hours
  Area under the concentration-time curve from time zero until the last observed concentration under fed conditions
Calculation of AUC0-inf for CRS3123 under fasted conditions | 24 hours
  Area under the concentration-time curve from time zero to infinity (extrapolated) under fasted conditions
Calculation of AUC0-inf for CRS3123 under fed conditions | 24 hours
  Area under the concentration-time curve from time zero to infinity (extrapolated) under fed conditions
Calculation of Cmax for CRS3123 under fasted conditions | 24 hours
  Maximal observed concentration under fasted conditions
Calculation of Cmax for CRS3123 under fed conditions | 24 hours
  Maximal observed concentration under fed conditions

SECONDARY OUTCOMES:
Calculation of Tmax for CRS3123 under fasted conditions | 24 hours
  Time when the maximal concentration is observed under fasted conditions
Calculation of Tmax for CRS3123 under fed conditions | 24 hours
  Time when the maximal concentration is observed under fed conditions
Calculation of Tlag for CRS3123 under fasted conditions | 24 hours
  Time of observation prior to the first observation with a measurable (non-zero) concentration under fasted conditions
Calculation of Tlag for CRS3123 under fed conditions | 24 hours
  Time of observation prior to the first observation with a measurable (non-zero) concentration fed conditions
Calculation of t1/2 for CRS3123 under fasted conditions | 24 hours
  Terminal elimination half-life under fasted conditions
Calculation of t1/2 for CRS3123 under fed conditions | 24 hours
  Terminal elimination half-life under fed conditions
Calculation of Kel for CRS3123 under fasted conditions | 24 hours
  Terminal elimination rate constant under fasted conditions
Calculation of Kel for CRS3123 under fed conditions | 24 hours
  Terminal elimination rate constant under fed conditions
Calculation of Cl/F for CRS3123 under fasted conditions | 24 hours
  Apparent clearance under fasted conditions
Calculation of Cl/F for CRS3123 under fed conditions | 24 hours
  Apparent clearance under fed conditions
Calculation of Vz/F for CRS3123 under fasted conditions | 24 hours
  Apparent volume of distribution under fasted conditions
Calculation of Vz/F for CRS3123 under fed conditions | 24 hours
  Apparent volume of distribution under fed conditions
Calculation of Tmax for CRS3123-glu3 metabolite under fasted conditions | 24 hours
  Time when the maximal concentration is observed under fasted conditions
Calculation of Tmax for CRS3123-glu3 metabolite under fed conditions | 24 hours
  Time when the maximal concentration is observed under fed conditions
Calculation of Tlag for CRS3123-glu3 metabolite under fasted conditions | 24 hours
  Time of observation prior to the first observation with a measurable (non-zero) concentration under fasted conditions
Calculation of Tlag for CRS3123-glu3 metabolite under fed conditions | 24 hours
  Time of observation prior to the first observation with a measurable (non-zero) concentration under fed conditions
Calculation of t1/2 for CRS3123-glu3 metabolite under fasted conditions | 24 hours
  Terminal elimination half-life under fasted conditions
Calculation of t1/2 for CRS3123-glu3 metabolite under fed conditions | 24 hours
  Terminal elimination half-life under fed conditions
Calculation of Kel for CRS3123-glu3 metabolite under fasted conditions | 24 hours
  Terminal elimination rate constant under fasted conditions
Calculation of Kel for CRS3123-glu3 metabolite under fed conditions | 24 hours
  Terminal elimination rate constant under fed conditions

CONTACTS AND LOCATIONS:
Locations (1):
- Syneos Health Miami, Miami, Florida, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT06988423/ICF_000.pdf